CLINICAL TRIAL: NCT02207725
Title: A Phase 3 Randomized, Double-Blind, Placebo-controlled Study in Older Subjects to Assess Safety and the Reversal of Apixaban Anticoagulation With Intravenously Administered Andexanet Alfa
Brief Title: A Study in Older Subjects to Evaluate the Safety and Ability of Andexanet Alfa to Reverse the Anticoagulation Effect of Apixaban
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Portola Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Alexion Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-503
Record Dates: First submitted 2014-04-28; First posted 2014-08-04 (Estimated); Results first posted 2018-09-27 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Bleeding
Keywords: Andexanet alpha; Anticoagulation; Antidote; Apixaban; Anti-fXa inhibitor; PRT4445; Eliquis; Reversal agent
MeSH Terms: conditions — Hemorrhage | interventions — PRT064445

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Andexanet (Experimental): Andexanet (antidote)
  Interventions: Biological: Andexanet
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Andexanet
  Arms: Andexanet
Other: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this stuy is to evaluate the ability of Andexanet Alfa to reverse the anticoagulation effect of Apixaban.

ELIGIBILITY:
Inclusion Criteria:

* Reasonably healthy men and women aged 50 to 75

Exclusion Criteria:

* History of abnormal bleeding, active bleeding or risk factors for bleeding
* History of thrombosis or risk factors for thrombosis
* History of adult asthma or use of inhaled medications

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2014-03; Primary Completion 2015-04 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vandana Mathur, M.D., Study Director — Portola Pharmaceuticals
Locations (1):
- Celerion, Tempe, Arizona, United States

REFERENCES:
- [Derived] Siegal DM, Curnutte JT, Connolly SJ, Lu G, Conley PB, Wiens BL, Mathur VS, Castillo J, Bronson MD, Leeds JM, Mar FA, Gold A, Crowther MA. Andexanet Alfa for the Reversal of Factor Xa Inhibitor Activity. N Engl J Med. 2015 Dec 17;373(25):2413-24. doi: 10.1056/NEJMoa1510991. Epub 2015 Nov 11. PMID 26559317

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject recruitment occurred at investigative site in the US between March 2014 through December 2014
Pre-assignment Details: Apixaban was administered orally at 5 mg twice daily for 3.5 days to steady-state and then administered andexanet as a bolus (400 mg; Part I) or as a bolus followed by an infusion (400 mg bolus followed by 4 mg/min infusion for 120 minutes, 880 mg total dose; Part II). Bolus was started 3 hours after the last apixaban dose.
Groups:
- Placebo (Part I): Placebo was administered intravenously (IV) as a bolus (Part I). The bolus was started 3 hours after the last apixaban dose (at the approximate steady-state Cmax for apixaban).
- Andexanet (Part I): Andexanet was administered IV as a bolus of 400 mg at a target rate of approximately 30 mg/minute (Part I). The bolus was started 3 hours after the last apixaban dose (at the approximate steady-state Cmax for apixaban)
- Placebo (Part II): Placebo was administered IV as a bolus followed by a continuous infusion for 120 minutes (Part II). The bolus was started 3 hours after the last apixaban dose (at the approximate steady-state Cmax for apixaban).
- Andexanet (Part II): Andexanet was administered IV as a bolus of 400 mg at a target rate of approximately 30 mg/minute, followed by a continuous infusion of 480 mg at 4 mg/minute for 120 minutes (Part II). The bolus was started 3 hours after the last apixaban dose (at the approximate steady-state Cmax for apixaban)
Period: Overall Study
Arm/Group | Placebo (Part I) | Andexanet (Part I) | Placebo (Part II) | Andexanet (Part II)
Started | 9 | 25 | 9 | 25
Completed | 9 | 24 | 8 | 24
Not Completed | 0 | 1 | 1 | 1
Not completed — Did Not Receive Treatment | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: 33 and 32 subjects were randomized in Part I and Part II of study, respectively
Groups:
- Andexanet (Part I): Andexanet was administered IV as a bolus of 400 mg at a target rate of approximately 30 mg/minute (Part 1). The bolus was started 3 hours after the last apixaban dose (at the approximate steady-state Cmax for apixaban)
- Total: Total of all reporting groups
Arm/Group | Placebo (Part I) | Andexanet (Part I) | Placebo (Part II) | Andexanet (Part II) | Total
Number analyzed (Participants) | 9 | 24 | 8 | 24 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (3.54) | 61.0 (6.37) | 59.5 (6.91) | 59.4 (7.83) | 59.9 (6.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 11 | 3 | 7 | 24
  Male | 6 | 13 | 5 | 17 | 41

OUTCOME MEASURES:

1. Primary Outcome: Efficacy: Percent Change From Baseline in Anti-fXa Activity at the Nadir (Parts I and II)
Description: In Part I, the primary endpoint was percent change from baseline in anti-fXa activity at the nadir, when nadir was defined as the smaller value for anti-fXa activity at the +2 minutes or +5 minutes time point following the end of the bolus. In Part II, the primary endpoint was the percent change from baseline in anti-fXa activity from its baseline to nadir, when nadir was defined as the smaller value for anti-fXa activity between the 110-minute time point (10 minutes prior to the end of the continuous infusion) and the 5-minute time point after the end of the continuous infusion. The baseline for the primary endpoint in both parts was the anti-fXa activity just prior to administration of andexanet, 3 hours following the Day 4 dose of apixaban. Anti-fXa activity was measured by a modified chromogenic assay.
Time Frame: Baseline to +2 minutes or +5 minutes following the end of andexanet/placebo bolus (Part I), or 10 minutes prior to end of andexanet/placebo continuous infusion or 5 minutes after the end of andexanet/placebo continuous infusion (Part II)
Population: Modified Intent-to-Treat Population included all subjects receiving andexanet/placebo with anti-fXa activity baseline value at ≥1 timepoints: 2 or 5 minute after the end of the bolus (Part I; N = 33); 110 minute during continuous infusion, 2 minute before or 5 minute after the end of continuous infusion (Part II; N = 31).
Measure: Mean (Standard Deviation); unit: Percent change in anti-fXa activity
Arm/Group | Placebo (Part I) | Andexanet (Part I) | Placebo (Part II) | Andexanet (Part II)
Number analyzed (Participants) | 9 | 24 | 8 | 23
Percent change in anti-fXa activity | -20.71 (8.559) | -93.86 (1.650) | -32.70 (5.578) | -92.34 (2.809)
Statistical Analysis 1: Comparison: Placebo (Part I) vs Andexanet (Part I); Test type: Superiority; p < 0.0001, 2-sided test exact Wilcoxon rank-sum tes; Hodges-Lehman estimate of shift = -74.55, 95% CI 2-sided [-78.39 to -66.28]
Statistical Analysis 2: Comparison: Placebo (Part II) vs Andexanet (Part II); Test type: Superiority; p < 0.0001, 2-sided test exact Wilcoxon rank-sum tes; Hodges-Lehman estimate of shift = -59.50, 95% CI 2-sided [-64.10 to -55.17]

2. Secondary Outcome: Efficacy: Percent Change From Baseline in Anti-fXa Activity at the Nadir (Part II)
Description: The percent change from baseline in anti-fXa activity at the nadir, following the bolus, when nadir was defined as the smaller value for anti-fXa activity at the +2 minute or +5 minute time point after the completion of the andexanet bolus (Part II). Baseline was the last assessment obtained prior to the first dose of andexanet or placebo
Time Frame: Baseline to +2 minutes or +5 minutes following the end of andexanet/placebo bolus (Part II)
Population: mITT; 33 and 31 subjects who received andexanet or placebo were included in the PD analysis in Part I and II, respectively.
Measure: Mean (Standard Deviation); unit: Percent change in anti-fXa activity
Arm/Group | Placebo (Part II) | Andexanet (Part II)
Number analyzed (Participants) | 8 | 23
Percent change in anti-fXa activity | -16.73 (4.104) | -93.49 (1.525)
Statistical Analysis 1: Comparison: Placebo (Part II) vs Andexanet (Part II); Test type: Superiority; p < 0.0001, 2-sided test exact Wilcoxon rank-sum tes; Hodges-Lehman estimate of shift = -77.14, 95% CI 2-sided [-79.98 to -74.04]

3. Secondary Outcome: Efficacy: Number of Participants With ≥80% Reduction in the Anti-fXa Activity From Baseline to Nadir
Description: Occurrence of ≥80% reduction in anti-fXa activity from its baseline to nadir, when nadir was defined as the smaller value for anti-fXa activity at the +2 minute or +5 minute time point after the completion of the andexanet bolus (Part I) or between the 110-minute time point (10 minutes prior to the end of the continuous infusion) and the 5-minute time point after the end of the continuous infusion (inclusive) [Part II]. Baseline was the last assessment obtained prior to the first dose of andexanet or placebo
Time Frame: as for outcome 1
Population: mITT; 33 and 31 subjects who received andexanet or placebo were included in the pharmacodynamics (PD) analysis in Part I and II, respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Part I) | Andexanet (Part I) | Placebo (Part II) | Andexanet (Part II)
Number analyzed (Participants) | 9 | 24 | 8 | 23
Participants | 0 | 24 | 0 | 23

4. Secondary Outcome: Efficacy -Change From Baseline in Free Apixaban Concentration at the Nadir
Description: Change from baseline in free apixaban concentration (ng/mL) at the nadir, when nadir was defined as the smaller value for free apixaban at the +2 minute or +5 minute time point after the completion of the andexanet bolus (Part I) or between the 110-minute time point (10 minutes prior to the end of the continuous infusion) and the 5-minute time point after the end of the continuous infusion (inclusive) [Part II]. Free plasma concentrations of apixaban was determined using a validated method that involved analysis of citrated human plasma with high-throughput equilibrium dialysis followed by liquid chromatography mass spectrometry.
Time Frame: as for outcome 1
Population: 54 subjects who received apixaban were included in the apixaban pharmacokinetics (PK) analysis
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo (Part I) | Andexanet (Part I) | Placebo (Part II) | Andexanet (Part II)
Number analyzed (Participants) | 9 | 24 | 8 | 23
ng/mL | -1.854 (1.6152) | -9.338 (3.2043) | -2.964 (1.1567) | -6.480 (2.7814)
Statistical Analysis 1: Comparison: Placebo (Part I) vs Andexanet (Part I); Test type: Superiority; p < 0.0001, 2-sided test exact Wilcoxon rank-sum tes; Hodges-Lehman estimate of shift = -7.09, 95% CI 2-sided [-8.86 to -5.42]
Statistical Analysis 2: Comparison: Placebo (Part II) vs Andexanet (Part II); Test type: Superiority; p = 0.0002, 2-sided test exact Wilcoxon rank-sum tes; Hodges-Lehman estimate of shift = -3.02, 95% CI 2-sided [-5.66 to -1.25]

5. Secondary Outcome: Efficacy: Change in Thrombin Generation (ETP) From Baseline to Its Peak [Parts I and II]
Description: Change in ETP from baseline to its peak, where peak was defined as the largest value for ETP between the +2 minute time point and the +10 minute time point after the end of the andexanet bolus (inclusive) {Part I] or between the 110-minute time point (10 minutes prior to the end of the continuous infusion) and the 5-minute time point after the end of the continuous infusion (inclusive) [Part II]. Baseline was the last assessment obtained prior to the first dose of andexanet or placebo. ETP was measured using a tissue factor-initiated thrombin generation assay.
Time Frame: Baseline to +2 minutes or +10 minutes following the end of andexanet/placebo bolus (Part I), or 10 minutes prior to end of andexanet/placebo continuous infusion or 5 minutes after the end of andexanet/placebo continuous infusion (Part II)
Population: 33 and 31 subjects who received andexanet or placebo were included in the PD analysis in Part I and II, respectively; mITT population
Measure: Mean (Standard Deviation); unit: nmol/min
Arm/Group | Placebo (Part I) | Andexanet (Part I) | Placebo (Part II) | Andexanet (Part II)
Number analyzed (Participants) | 9 | 24 | 8 | 23
nmol/min | 88.182 (125.7621) | 1323.180 (335.4321) | 189.409 (184.7842) | 1193.060 (263.3471)
Statistical Analysis 1: Comparison: Placebo (Part I) vs Andexanet (Part I); Test type: Superiority; p < 0.0001, 2-sided test exact Wilcoxon rank-sum tes; Hodges-Lehman estimate of shift = 1227.35, 95% CI 2-sided [984.01 to 1456.38]
Statistical Analysis 2: Comparison: Placebo (Part II) vs Andexanet (Part II); Test type: Superiority; p < 0.0001, 2-sided test exact Wilcoxon rank-sum tes; Hodges-Lehman estimate of shift = 999.33, 95% CI 2-sided [819.50 to 1200.53]

6. Secondary Outcome: Efficacy: Number of Participants With Thrombin Generation (ETP) Above the Lower Limit of the Derived Normal Range at Its Peak (mITT Population)
Description: Number of participants with ETP above the lower limit of the normal range at its peak, between the +2 minute time point and the +10 minute time point after the end of the andexanet bolus (inclusive) [Part I] or between the 110-minute time point (10 minutes prior to the end of the continuous infusion) and the 5-minute time point after the end of the continuous infusion (inclusive) [Part II]. ETP was measured using a tissue factor-initiated thrombin generation assay
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Part I) | Andexanet (Part I) | Placebo (Part II) | Andexanet (Part II)
Number analyzed (Participants) | 9 | 24 | 8 | 23
Participants | 1 | 24 | 2 | 23

ADVERSE EVENTS:
Time Frame: ~8 to 12 weeks
Description: The Safety Analysis Population consisted of all subjects randomized and treated with study drug (andexanet or placebo)
Groups:
- Placebo (Part I); Placebo (Part II): Vehicle Control
- Andexanet (Part I): 400 mg bolus
- Andexanet (Part II): 400 mg bolus + 480 mg infusion (4 mg/min)
Arm/Group | Placebo (Part I) | Andexanet (Part I) | Placebo (Part II) | Andexanet (Part II)
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/24 | 0/8 | 0/24
Other Adverse Events (participants affected / at risk) | 3/9 | 7/24 | 2/8 | 9/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Part I) (N=9) | Andexanet (Part I) (N=24) | Placebo (Part II) (N=8) | Andexanet (Part II) (N=24)
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Vessel Puncture Site Haemorrhage (General disorders) | 1 | 0 | 0 | 4
Vessel Puncture Site Pain (General disorders) | 1 | 2 | 0 | 0
Vessel Puncture Site Swelling (General disorders) | 0 | 0 | 0 | 2
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 3 | 2 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Headache (Nervous system disorders) | 1 | 3 | 0 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 | 3 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Conducted in healthy volunteers at Clinical Research Organization.